CLINICAL TRIAL: NCT05968378
Title: Immunometabolic Effects of Time Restricted Eating in Non-alcoholic Fatty Liver Disease
Brief Title: Diet, Immunometabolism and Non-alcoholic Fatty Liver Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College Dublin (Other)
Collaborators: St. James's Hospital, Ireland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LS-E-22-105-Shannon-Roche
Record Dates: First submitted 2023-06-26; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Liver Fat; Obesity; Inflammation
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Obesity; Inflammation | interventions — Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard healthy eating advice (Active Comparator): Subjects in this group will be counselled according to the Irish National Healthy Eating Guidelines.
  Interventions: Behavioral: Standard healthy eating advice
- eTRE plus Mediterranean diet (Experimental): Subjects in this group will be asked to restrict their eating to 8-hours daily (8am - 4pm) and to adhere to a Mediterranean style diet.
  Interventions: Behavioral: eTRE plus Mediterranean diet

INTERVENTIONS:
Behavioral: Standard healthy eating advice — Subjects in this group will be provided with standard healthy eating advice according to the Irish National Healthy Eating Guidelines and Food Pyramid and will be asked to follow this advice for 8-weeks.
  Arms: Standard healthy eating advice
Behavioral: eTRE plus Mediterranean diet — Subjects in this group will be asked to consume all meals between 8am - 4pm and to adhere to a Mediterranean style diet daily for 8-weeks.
  Arms: eTRE plus Mediterranean diet

SUMMARY:
This study will assess the impact of 8-hour time restricted eating (8 hours of eating, 16 hours fasting) combined with a Mediterranean diet on metabolism and inflammation in adults with non-alcoholic fatty liver disease (NAFLD).

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD), defined as the accumulation of fat in the liver that is not related to alcohol intake, is the number 1 global cause of chronic liver disease. Excessive consumption of energy, saturated fat, and simple sugars is a key contributor to hepatic lipid accumulation and obesity-induced metabolic inflammation, reflecting cross-talk between immune and metabolic pathways. Moreover, dietary factors including saturated fatty acids, cholesterol, and their derivatives, as well as gut-derived metabolites, can prime innate immune cells to induce an exaggerated pro-inflammatory response upon re-exposure to such stimuli and may contribute to chronic low grade inflammation.

Dietary strategies focusing on replacing inflammatory dietary triggers with monounsaturated fats, fiber and complex carbohydrates have been shown to improve metabolic dysfunction, but how this relates to a rewiring of the innate immune system is less clear. Time-restricted eating (TRE) is another dietary strategy which has been shown to elicit beneficial effects that reduce the risk of chronic metabolic disease and consolidates eating to a 6-10 hour period daily. Early TRE (eTRE), wherein eating occurs from morning to early afternoon, is associated with greater cardiometabolic health benefits than eating late in the evening. This includes improved insulin sensitivity, glucose tolerance and lipid metabolism, and reduced inflammatory markers.

This study will determine the impact of an 8-week intervention of 8-hour eTRE combined with an anti-inflammatory Mediterranean diet on the metabolic and immune phenotype of individuals with NAFLD, a population at high risk of progressive cardiometabolic decline and chronic inflammation. By focusing on improving both nutrient quality and nutrient timing, a greater understanding of the interaction between systemic metabolism and immune cell rewiring will be gained.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Age 18-65 years, from all ethnic groups, capable of providing informed consent to participate
* Obesity (body mass index >30kg/m^2) and of stable body weight (±3% for ≥3 months)
* Fasting blood glucose <7.0 mmol/L and HbA1c <6.5%.
* Liver fat >10% (CAP score >238 dB/m) and no fibrosis (liver stiffness score 2-7 kPa) as assessed by liver elastography (FibroScan)

Exclusion Criteria:

* Impaired renal function
* Abnormal hematocrit
* History of cardiovascular events
* Uncontrolled hypertension
* Type 2 diabetes
* Medications or supplements known to affect glucose or lipid metabolism
* Active inflammatory, autoimmune, infectious, gastrointestinal, or malignant disease
* Uncontrolled neurological or psychiatric disease
* Iron deficiency anemia, (hemoglobin < 12g/dl men, < 11g/dl women)
* Fatty acid supplements and consumers of high doses of anti- antioxidant vitamins (A, C, E, b-carotene)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Change in plasma inflammatory response to a high-fat meal: C-reactive protein (CRP) | To be assessed at baseline and post 8-week intervention
  Postprandial changes in CRP (mg/L) will be measured in response to a high-fat meal
Change in plasma inflammatory response to a high-fat meal: Interleukin-6 (IL-6) | To be assessed at baseline and post 8-week intervention
  Postprandial changes in IL-6 (pg/mL) will be measured in response to a high-fat meal
Change in plasma inflammatory response to a high-fat meal: Interleukin-1-beta (IL-1β) | To be assessed at baseline and post 8-week intervention
  Postprandial changes in IL-1β (pg/mL) will be measured in response to a high-fat meal
Change in plasma inflammatory response to a high-fat meal: Tumor necrosis factor alpha (TNF-α) | To be assessed at baseline and post 8-week intervention
  Postprandial changes in (TNF-α) (pg/mL) will be measured in response to a high-fat meal

SECONDARY OUTCOMES:
Change in metabolic response to a high-fat meal: Glucose | To be assessed at baseline and post 8-week intervention
  Plasma glucose (mg/dL) response to a high-fat meal will be assessed
Change in metabolic response to a high-fat meal: Insulin | To be assessed at baseline and post 8-week intervention
  Plasma insulin (μU/mL) response to a high-fat meal will be assessed
Change in metabolic response to a high-fat meal: Glucagon | To be assessed at baseline and post 8-week intervention
  Plasma glucagon (pg/mL) response to a high-fat meal will be assessed
Change in metabolic response to a high-fat meal: Triglycerides | To be assessed at baseline and post 8-week intervention
  Plasma triglycerides (mg/dL) response to a high-fat meal will be assessed
Change in metabolic response to a high-fat meal: Non-esterified fatty acids (NEFA) | To be assessed at baseline and post 8-week intervention
  Plasma NEFA (mmol/L) response to a high-fat meal will be assessed
Innate immune function | To be assessed at baseline and post 8-week intervention
  8-week change in innate immune function will be assessed ex-vivo using whole blood simulation assay.
Innate immune training | To be assessed at baseline and post 8-week intervention
  8-week change in innate immune function will be assessed in isolated monocytes stimulated with beta glucan and restimulated with lipopolysaccharide.
Insulin resistance | To be assessed at baseline and post 8-week intervention
  8-week change in insulin resistance using Homeostatic Model Assessment for Insulin Resistance (HOMA-IR).
Adipose tissue insulin resistance | To be assessed at baseline and post 8-week intervention
  8-week change in adipose tissue insulin resistance using the adipose tissue insulin resistance index (Adipo-IR).
Change in intrahepatic triglyceride content | To be assessed at baseline and post 8-week intervention
  Liver elastography (FibroScan) will be used to determine change in liver fat after the 8-week intervention.
Change in liver stiffness measurement | To be assessed at baseline and post 8-week intervention
  Liver elastography (FibroScan) will be used to determine change in liver stiffness after the 8-week intervention.
HDL Proteome | To be assessed at baseline and post 8-week intervention
  8-week change in the composition of the HDL proteome.
Body weight | To be assessed at baseline and post 8-week intervention
  8-week change in body weight in kilograms
Body mass index (BMI) | To be assessed at baseline and post 8-week intervention
  8-week change in BMI
Body fat percentage | To be assessed at baseline and post 8-week intervention
  8 week change in body fat percentage using bioelectrical impedance analysis
Waist and hip circumferences | To be assessed at baseline and post 8-week intervention
  8-week change in waist and hip circumference measured in centimeters using a body tape measure
Gut microbiome composition and function | To be assessed at baseline and post 8-week intervention
  8-week functional changes in gut microbiome will be assessed by integrating 16S sequencing of fecal samples with fecal water metabolomics.
Dietary intake | To be assessed at baseline and post 8-week intervention
  8-week change in dietary intake using a 3-day semi-weighed food diary.
Physical activity level (PAL) | To be assessed at baseline and post 8-week intervention
  8-week change in PAL using the International Physical Activity Questionnaire - Short form (IPAQ-SF). This form has 7 questions about time spent doing physical activity(leisure time, work, domestic tasks, and travel) in the last 7 days. Activities are grouped according to vigorous or moderate intensity, and walking. Each intensity is assigned a metabolic equivalent (MET). The time spent at each intensity is used to estimate weekly physical activity using the associated METs. Minimum and maximum values are 0 and 154,224 METs. Classification as 'sufficiently active' requires ≥600 METs/week which may be achieved through a combination of intensities. Classification as 'highly active' requires: a) vigorous-intensity activity on ≥3 days achieving a minimum of ≥1500 METs/week OR b) ≥7 days of any combination of walking, moderate-intensity or vigorous-intensity activities achieving ≥ 3000 METs/week. A physical activity level below these categories is undesirable.
Mediterranean diet adherence | To be assessed at baseline and post 8-week intervention
  8-week change in Mediterranean diet adherence score using the PREDIMED 14-item Mediterranean Diet Assessment Tool. This questionnaire is used to assess adherence to the traditional Mediterranean Diet. Two of the 14 questions relate to the use of olive oil, a key component of the Mediterranean Diet, and 12 questions relate to the consumption of foods which characterize the Mediterranean Diet. Each item has a criteria which must be met to achieve 1 point e.g., at least 3 pieces of fruit daily. The minimum score is 0 and the maximum is 14, where a score of ≤ 5 indicates low adherence, 6-9 moderate adherence, and > 9 high adherence.

CONTACTS AND LOCATIONS:
Locations (1):
- University College Dublin, Dublin, Leinster, Ireland